CLINICAL TRIAL: NCT03904914
Title: Development of a New Simplified Thumb Ossification Composite Index (TOCI) and Its Application to Predict Skeletal Maturity and Curve Progression in Idiopathic Scoliosis and Normal Subjects
Brief Title: Thumb Ossification Composite Index (TOCI) to Predict Skeletal Maturity and Curve Progression in AIS
Acronym: TOCI
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Alec Lik-Hang Hung, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: 2016.045
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Scoliosis; Adolescence; Bone Diseases; Bone Growth Abnormal
Keywords: TOCI; scoliosis
MeSH Terms: conditions — Scoliosis; Bone Diseases; Bone Diseases, Developmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIS group: Patients confirmed with adolescent idiopathic scoliosis (AIS)
  Interventions: Other: TOCI

INTERVENTIONS:
Other: TOCI — TOCI staging evaluated

SUMMARY:
Accurate skeletal maturity assessment is important for prediction of curve progression and clinical management of adolescent idiopathic scoliosis (AIS) including bracing decision and counseling for prognosis. Determination of the timing of peak growth height velocity and growth remaining are paramount important.1,2 Commonly used clinical or radiological methods are still inadequate or too complex for rapid clinical use in the outpatient setting.3-5 Risser sign had disadvantages of low visibility in posteroanterior (PA) spinal radiograph, wide variability with maturity level and imprecise representation of peak height velocity (PHV) timing.6 Greulich and Pyle atlas (GP atlas) and Tanner-Whitehouse-III (TWIII) method are more reliable and comprehensive classifications to predict maturity, but they are cumbersome and time consuming to be used clinically.7 Both methods require the usage of an atlas, a learning curve required for exact matching of atlas plate or assignment of scores to bones.8

In this study, the investigators introduce Thumb Ossification Classification Index (TOCI). TOCI employed the measurements of epiphysis of distal phalange, proximal phalange, and adductor sesamoid, and results were analyzed together to form a composite stage (composite score) to predict maturity in patient at their peripubertal period. Ultimately the application of TOCI should not be limited to IS patients only. After the establishment of TOCI classification system, the staging system would be applied to radiographs from patients without spinal deformity or suffering from diseases not related to spine.

DETAILED DESCRIPTION:
Introduction

Accurate skeletal maturity assessment is important for prediction of curve progression and clinical management of adolescent idiopathic scoliosis (AIS) including bracing decision and counseling for prognosis. Determination of the timing of peak growth height velocity and growth remaining are paramount important.1,2 Commonly used clinical or radiological methods are still inadequate or too complex for rapid clinical use in the outpatient setting.3-5 Risser sign had disadvantages of low visibility in PA spinal radiograph, wide variability with maturity level and imprecise representation of PHV timing.6 Greulich and Pyle atlas (GP atlas) and Tanner-Whitehouse-III (TWIII) method are more reliable and comprehensive classifications to predict maturity, but they are cumbersome and time consuming to be used clinically.7 Both methods require the usage of an atlas, a learning curve required for exact matching of atlas plate or assignment of scores to bones.8

Some latest skeletal maturity bone models were evolved trying to solve these problems but were still imperfect.9 Recently, Sanders made modifications to TWIII method to form Skeletal Maturity Scoring System (SMSS) which focused on epiphysis of small hand bones from all 5 digits. SMSS was proved to have excellent correlation with the curve acceleration phase.10 Digital skeletal age scores between 400 and 425 are associated with the beginning of the curve acceleration phase in adolescent idiopathic scoliosis.11 Excellent intra-observer reliability and substantial inter-observer reliability among senior surgeons were demonstrated in SMSS.12

A new skeletal age classification has yet to be developed, although SMSS has considered a promising method. A recent study to test SMSS's reliability in less experienced staffs demonstrated average inter-observer reliability (K=0.53).8 It showed that a learning curve was present and several recommendations were added in each classification stage to avoid controversy and confusion during usage.13 Therefore, using SMSS requires an organized teaching system with detailed descriptions, self-assessment examinations, viewing presentations and the newly added recommended modification guidelines to improve the reliability. Another scoring system "Distal Radius and Ulna (DRU)" score simplified the measurement to just using radial and ulnar epiphyses but results observed that DRU score had the least correlation of "Radio Ulna and Short bones" (RUS) growth centers with scoliosis behavior.9,10 In addition, the variable appearance of ulnar epiphysis were difficult to be seen clearly.

In this study, the investigators introduce Thumb Ossification Classification Index (TOCI). TOCI employed the measurements of epiphysis of distal phalange, proximal phalange, and adductor sesamoid, and results were analyzed together to form a composite stage (composite score) to predict maturity in patient at their peripubertal period. Ultimately the application of TOCI should not be limited to IS patients only. After the establishment of TOCI classification system, the staging system would be applied to radiographs from patients without spinal deformity or suffering from diseases not related to spine.

The objectives of this study were as follows:

1. Measure different bony features at hand bones and classify the bony features to TOCI stages
2. Evaluate the TOCI system by comparing the measured TOCI stages with digital skeletal age (DSA) and radio ulna and short bones (RUS) scores
3. Evaluate the intra-rater and inter-rater reliability of TOCI system

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Pre-menarche
* Confirmed diagnosis of idiopathic scoliosis
* No evidence of neurological abnormality
* No abnormalities of maturation
* Risser sign of zero in spinal radiograph and open physis in hand radiograph

Exclusion Criteria:

* Patients with diagnosis of non-idiopathic scoliosis, e.g. congenital, neuromuscular , syndromal cause of scoliosis
* Patients with maturation abnormality (either precocious puberty or developmental delay)
* Abnormalities of the head or neck that would change height measurements
* Previous history of spinal fusion operation performed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Scoliosis patients will be recruited from a specialized scoliosis clinic in Prince of Wales hospital visiting the clinic.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TOCI stage | Baseline, from X-ray scans, higher values represent more mature bone
  Evaluate TOCI stage from 1 to 8

CONTACTS AND LOCATIONS:
Overall Officials: Alec Lik-Hang Hung, Dr., Principal Investigator — Department of Orthopaedics and Traumatology, Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hung ALH, Chau WW, Shi B, Chow SK, Yu FYP, Lam TP, Ng BKW, Qiu Y, Cheng JCY. Thumb Ossification Composite Index (TOCI) for Predicting Peripubertal Skeletal Maturity and Peak Height Velocity in Idiopathic Scoliosis: A Validation Study of Premenarchal Girls with Adolescent Idiopathic Scoliosis Followed Longitudinally Until Skeletal Maturity. J Bone Joint Surg Am. 2017 Sep 6;99(17):1438-1446. doi: 10.2106/JBJS.16.01078. PMID 28872525
- [Result] Hung AL, Shi B, Chow SK, Chau WW, Hung VW, Wong RM, Liu KL, Lam TP, Ng BK, Cheng JC. Validation Study of the Thumb Ossification Composite Index (TOCI) in Idiopathic Scoliosis: A Stage-to-Stage Correlation with Classic Tanner-Whitehouse and Sanders Simplified Skeletal Maturity Systems. J Bone Joint Surg Am. 2018 Jul 5;100(13):88. doi: 10.2106/JBJS.17.01271. PMID 29975274